CLINICAL TRIAL: NCT03220672
Title: Effectiveness of a Tailored Assessment and Educational Intervention on Motor Control of the Pelvic Floor Muscle in Menopausal and Peri-menopausal Women
Brief Title: Effectiveness of Assessment and Educational Intervention on Motor Control of the Pelvic Floor Muscle in Women
Acronym: MENO_edu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Principal Researcher of CTS631 University of Malaga, University of Malaga
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Meno_Edu_2017
Record Dates: First submitted 2017-07-04; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-06

CONDITIONS: Menopause; Perimenopausal Disorder
Keywords: Pelvic floor muscles; pelvic floor muscle training; motor control; Educational intervention; menopause

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Expertimental (Experimental): The sample will receive a tailored assessment and educational intervention on Motor Control of the Pelvic Floor Muscle
  Interventions: Behavioral: Tailored assessment and educational

INTERVENTIONS:
Behavioral: Tailored assessment and educational — Intervention will consist of 45 minutes of anatomy education, pelvic floor assessment and neuromuscular re-education. Women will be given an explanation of how the pelvis is composed, including the viscera and pelvic floor function and anatomy, through a simple explanatory sheet. They will be also informed of the causes of pelvic floor deterioration as well as its consequences.. Neuromuscular re-education will continued by teaching them how to perform slow contractions, fast contractions and lifting contraction. They will be also shown vaginal cones and advised on possible treatment methods if they were needed. After that, women will be given a tip sheet to improve pelvic floor function. Those recommendations will included: Tips to take into account during habits like urination, doing sport, gymnastics or any efforts, pelvic floor muscles exercises and how to use vaginal cones adequately.

SUMMARY:
The goal of the present study is to evaluate the short and long term effectiveness of a tailored assessment and educational intervention on motor control of the pelvic floor muscle in menopausal and non-menopausal women.

DETAILED DESCRIPTION:
Menopausal transition has been related to stress urinary incontinence. The transition from the reproductive to the non-reproductive period is induced by a decrease in sex hormone production in the ovaries. Climacteric-stage oestrogen deficiency produces genital and urinary tract atrophy, which may be related to symptoms such as urinary frequency, urinary urgency, nocturia incontinence, and recurrent urinary tract infection. Urinary incontinence seems to appear due to a combination of factors such as pelvic floor weakness and tearing, denervation and fascial tears as well as both loss of motor units and altered activation patterns. However, physiotherapy can treat weakness and altered motor control in order to compensate for other factors. In fact, physiotherapy is considered the treatment of first choice.

Besides evidence defending physiotherapy as first line conservative therapy in incontinence due to influence of strength and motor control in this pathology and its prevalence in perimenopause women, little is known about its effects in this population. Hence, the aim of this study is to evaluate the short and long term effectiveness of a tailored assessment and educational intervention on motor control of the pelvic floor muscle in menopausal and peri-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* All participants in this study will sign an informed consent form prior their inclusion, and that whose participation will be voluntary

Exclusion Criteria:

* Participants will be excluded if they have any cognitive disability, physical disability or psychiatric limitations that could limit the participation on the study test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Due to the aim of the study, the gender of the sample will be female
Enrollment: 120 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Motor Control of Pelvic Floor Muscle by single questionnare | inmediate effect post education
  Women will report an outcome regarding tightening capacity after intervention. It consisted of a one item questionnaire about pelvic floor contraction capacity. It is chosen by the expert panel developed by researcher from this project. The item is a question regarding tightening capacity and it had a polychotomous answer:
  "How is the tightening capacity of your pelvic floor muscles?
  a) very high, b) high, c) good, d) optimal, e) bad, f) low, g) very low"

SECONDARY OUTCOMES:
Anthropometric | baseline, inmediate effect post education and 2,4 and 12 weeks. Long time effect 6 months
  Age, height and weight, and their Body Mass Index (BMI) was calculated.
Interview about urinary incontinence | baseline, inmediate effect post education and 2,4 and 12 weeks. Long time effect 6 months
  Women will also underwent an interview about urinary incontinence with a physiotherapist from the Consulting Unit of Physiotherapy of the Pelvic Floor. The questionnaire consisted of 38 items regarding delivery conditions, faecal and urinary incontinence as well as medical conditions and lifestyle. This interview includes information from descriptive outcomes reported by the clinician, so pelvic floor muscles will be evaluated by both manual muscle testing and a perineometer. Hence, this interview has both qualitative and quantitative reponses.
The International Consultation on Incontinence Questionnaire (ICIQ-UI SHORT FORM) | baseline, inmediate effect post education and 2,4 and 12 weeks. Long time effect 6 months
  The ICIQ is a simple and short questionnaire to assess the symptoms and impact of UI across the population. It consists of 3 items which indicate frequency, quantity and impact, and 8 questions more related to the symptoms indicative of the type of UI, but not being contemplated when obtaining a global index. The ICIQ-UI short form has a good reliability with a Cronbach's alpha of 0.95. It was validated in Spanish by Espuña et al, with a Cronbach's alpha of 0.89

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chevalier F, Fernandez-Lao C, Cuesta-Vargas AI. Normal reference values of strength in pelvic floor muscle of women: a descriptive and inferential study. BMC Womens Health. 2014 Nov 25;14:143. doi: 10.1186/s12905-014-0143-4. PMID 25420756
- [Background] Espuna Pons M, Rebollo Alvarez P, Puig Clota M. [Validation of the Spanish version of the International Consultation on Incontinence Questionnaire-Short Form. A questionnaire for assessing the urinary incontinence]. Med Clin (Barc). 2004 Mar 6;122(8):288-92. doi: 10.1016/s0025-7753(04)74212-8. Spanish. PMID 15030739
- [Background] Bo K. Pelvic floor muscle training is effective in treatment of female stress urinary incontinence, but how does it work? Int Urogynecol J Pelvic Floor Dysfunct. 2004 Mar-Apr;15(2):76-84. doi: 10.1007/s00192-004-1125-0. Epub 2004 Jan 24. PMID 15014933